CLINICAL TRIAL: NCT04091568
Title: Comparison of Patients' Experience Following Awake and Asleep Fibreoptic Intubation
Brief Title: Patient Experience Following Awake Fibreoptic Intubation Compared to Asleep Fibreoptic Intubation
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 247165
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Tracheal Intubation; Intubation;Difficult
Keywords: Awake fibre-optic tracheal intubation; Asleep fibre-optic tracheal intubation; Patient experience

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Awake fibre-optic intubation: Awake fibre-optic intubation
- Asleep fibre-optic intubation: Asleep fibre-optic intubation

SUMMARY:
The aim of this observational study is to explore and compare patients' experiences of asleep and awake fibreoptic intubation using a semi qualitative patient questionnaire. In particular, investigators will investigate the occurrence of negative experiences, such as distress and discomfort.

DETAILED DESCRIPTION:
This study aims to investigate whether there are significant differences in aspects of patient experience during AFOI and asleep fibreoptic intubation. The study will be conducted at University Hospitals Coventry and Warwickshire NHS Trust and Oxford University Hospitals Foundation Trust.

Investigators are not aware of any studies to date comparing patient experiences of AFOI with asleep fibreoptic intubation to ascertain the significant differences in side effects. If there is no evidence of any significant difference in negative patient experiences, this might help to encourage anaesthetists to reduce their threshold for AFOI and to use this as first choice for anticipated difficult airway management.

A member of the research team will approach the patient about the study and obtain written informed consent, if the patient is willing and able to participate. The participant will be provided with a specifically designed questionnaire, covering several aspects of patient experience. A mixture of free response answers and numerical rating scales will be used. The member of the research team approaching the patient with the questionnaire will be blinded to the intubation procedure, ensuring consistent application of the questionnaire and minimising bias. This will then be the end of the study for the participant.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 years and above
* Patients who underwent head and neck or dental surgery and required awake or asleep fibreoptic intubation
* Patients who underwent elective surgery
* Are able and willing to provide written informed consent

Exclusion Criteria:

* Patients who do not consent to be part of the study
* Patients below 18 years old If a translator is not available at the time, participants who cannot reasonably read and communicate in English
* Those who did not undergo awake or asleep fibreoptic intubation
* Those who underwent emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Those patients who undergo either awake or asleep fibreoptic intubation in the Head and Neck Theatres at both UHCW and Oxford University Hospitals Foundation Trust, as decided by their responsible anaesthetist.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
To assess the incidence and severity of distress experienced by patients during awake and asleep fibreoptic intubation. | 6 - 12 months
  Participants will be asked to rate the discomfort during the procedure on a Visual Analogue Score (0-10). There will also be space for patients to write comments explaining their score. These comments will then be used for content analysis, for example to explore different aspects of the procedure that caused distress.

SECONDARY OUTCOMES:
Secondary endpoints include the differences in occurrence of patient discomfort, pain and difficulty breathing. | 6 - 12 months
  This will be assessed through the patient experience questionnaire, with a mixture of direct questions and the request for more detailed information regarding these answers.

CONTACTS AND LOCATIONS:
Overall Officials: Ceri Jones, Study Chair — University Hospitals of Coventry and Warwickshire; Cyprian Mendonca, MD,FRCA, Principal Investigator — University Hospitals of Coventry and Warwickshire
Locations (2):
- United Kingdom (2):
  - University Hospitals Coventry & Warwickshire NHS Trust, Coventry, West Midlands
  - Oxford University Hospitals, Oxford

IPD SHARING:
Plan to Share IPD: No
IPD will be a written questionnaire which is anonymous

REFERENCES:
- [Background] Frerk C, Mitchell VS, McNarry AF, Mendonca C, Bhagrath R, Patel A, O'Sullivan EP, Woodall NM, Ahmad I; Difficult Airway Society intubation guidelines working group. Difficult Airway Society 2015 guidelines for management of unanticipated difficult intubation in adults. Br J Anaesth. 2015 Dec;115(6):827-48. doi: 10.1093/bja/aev371. Epub 2015 Nov 10. PMID 26556848
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Allan AG. Reluctance of anaesthetists to perform awake intubation. Anaesthesia. 2004 Apr;59(4):413. doi: 10.1111/j.1365-2044.2004.03729.x. No abstract available. PMID 15023129
- [Background] Patil V, Barker GL, Harwood RJ, Woodall NM. Training course in local anaesthesia of the airway and fibreoptic intubation using course delegates as subjects. Br J Anaesth. 2002 Oct;89(4):586-93. doi: 10.1093/bja/aef226. PMID 12393360
- [Background] Wanderer JP, Ehrenfeld JM, Sandberg WS, Epstein RH. The changing scope of difficult airway management. Can J Anaesth. 2013 Oct;60(10):1022-4. doi: 10.1007/s12630-013-9999-2. Epub 2013 Jul 30. No abstract available. PMID 23897492
- [Background] Wiles MD, McCahon RA, Armstrong JAM. Fibreoptic intubation rates in a UK teaching hospital. Proceedings of the Anaesthetic Research Society Meeting. Br J Anaesth 2010; 105 (5): 729P
- [Background] Heidegger T, Gerig HJ, Ulrich B, Kreienbuhl G. Validation of a simple algorithm for tracheal intubation: daily practice is the key to success in emergencies--an analysis of 13,248 intubations. Anesth Analg. 2001 Feb;92(2):517-22. doi: 10.1097/00000539-200102000-00044. PMID 11159261
- [Background] McNarry AF, Dovell T, Dancey FM, Pead ME. Perception of training needs and opportunities in advanced airway skills: a survey of British and Irish trainees. Eur J Anaesthesiol. 2007 Jun;24(6):498-504. doi: 10.1017/S0265021506002031. Epub 2007 Jan 8. PMID 17207298
- [Background] El-Boghdadly K, Onwochei DN, Cuddihy J, Ahmad I. A prospective cohort study of awake fibreoptic intubation practice at a tertiary centre. Anaesthesia. 2017 Jun;72(6):694-703. doi: 10.1111/anae.13844. PMID 28654138
- [Background] Mavridou P, Dimitriou V, Manataki A, Arnaoutoglou E, Papadopoulos G. Patient's anxiety and fear of anesthesia: effect of gender, age, education, and previous experience of anesthesia. A survey of 400 patients. J Anesth. 2013 Feb;27(1):104-8. doi: 10.1007/s00540-012-1460-0. Epub 2012 Aug 3. PMID 22864564
- [Background] Schnack DT, Kristensen MS, Rasmussen LS. Patients' experience of awake versus anaesthetised orotracheal intubation: a controlled study. Eur J Anaesthesiol. 2011 Jun;28(6):438-42. doi: 10.1097/EJA.0b013e328343222d. PMID 21544021
- [Background] Knudsen K, Nilsson U, Hogman M, Poder U. Awake intubation creates feelings of being in a vulnerable situation but cared for in safe hands: a qualitative study. BMC Anesthesiol. 2016 Aug 30;16(1):71. doi: 10.1186/s12871-016-0240-z. PMID 27576876